CLINICAL TRIAL: NCT00449410
Title: Silent Cerebrovascular Lesion and Cognitive Decline Prevention in Atrial Fibrillation by Intensive Cholesterol Lowering in Elderly Patients
Brief Title: Silent Cerebrovascular Lesion and Cognitive Decline Prevention by Cholesterol Lowering in Elderly AF Patients
Acronym: SPACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Pfizer (Industry); Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPACE1
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Atrial Fibrillation; Neuropsychology; Magnetic Resonance Imaging; Inflammation; Hemostasis
Keywords: Atrial Fibrillation; elderly; cholesterol lowering; neurocognitive function; cerebrovascular lesion
MeSH Terms: conditions — Atrial Fibrillation; Inflammation; Cerebrovascular Disorders | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atorvastatin
Drug: ezetimibe

SUMMARY:
In elderly patients with atrial fibrillation (AF) the presence of silent brain infarcts and neurocognitive deficit is high despite adequate treatment with oral anticoagulation. Atherosclerosis is considered to be a chronic inflammatory disease and thrombosis and inflammation are strongly correlated. Atrial fibrillation is linked with increased levels of inflammatory markers and intensive cholesterol lowering has proven to reduce inflammation. In a prospective double-blind randomized pilot-study we want to test the hypothesis, that addition of intensive cholesterol lowering treatment besides adequate oral anticoagulation will reduce cerebrovascular lesions and will be beneficial for neurocognitive status in elderly AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>68 and <82 years) with atrial fibrillation and adequate oral anticoagulation therapy and cholesterol levels between 4,5 mmol/l and 7 mmol/l

Exclusion Criteria:

* Indication for cholesterol lowering treatment according to Dutch CBO-cholesterol guidelines (2004)

Ages: 68 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35
Dates: Start 2005-05; Study Completion 2006-10

PRIMARY OUTCOMES:
Neurocognitive function
Cerebrovascular lesions on MRI

SECONDARY OUTCOMES:
Level of inflammatory markers
Level of hemostatic markers

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kuilenburg, MD, Principal Investigator — UMCN Radboud; Gheorghe AM Pop, MD PhD, Study Director — UMCN Radboud
Locations (1):
- Gheorghe AM Pop, Nijmegen, Netherlands

REFERENCES:
- [Derived] Lappegard KT, Pop-Purceleanu M, van Heerde W, Sexton J, Tendolkar I, Pop G. Improved neurocognitive functions correlate with reduced inflammatory burden in atrial fibrillation patients treated with intensive cholesterol lowering therapy. J Neuroinflammation. 2013 Jun 28;10:78. doi: 10.1186/1742-2094-10-78. PMID 23809138